CLINICAL TRIAL: NCT00828932
Title: An Open Label, Single Dose Study of the Pharmacokinetic Properties of Lorcaserin in Subjects With Hepatic Impairment
Brief Title: Pharmacokinetic Properties of Lorcaserin in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APD356-017
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-07

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorcaserin 10mg (Experimental)
  Interventions: Drug: Lorcaserin

INTERVENTIONS:
Drug: Lorcaserin

SUMMARY:
The purpose of this study is to evaluate and establish whether lorcaserin dose adjustment is required in patients with mild or moderate hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged between 18 and 75 years (inclusive)
2. Able to give signed informed consent
3. Hepatic function will fall into one of the following categories:

   * One-third of patients will have normal hepatic function (defined as having all of the following parameters within the normal range of the clinical laboratory used for this trial: AST, ALT, alkaline phosphatase, total bilirubin)
   * One-third of patients will have mild impairment (Child-Pugh score 5-6)
   * One-third of patients will have moderate impairment (Child-Pugh score 7-9)
4. All subjects will have a BMI of 27-45 kg/m2, inclusive.
5. Eligible male and female patients must agree not to participate in a conception process
6. Considered to be in stable health in the opinion of the Investigator.

Exclusion Criteria:

1. Prior participation in any study of lorcaserin.
2. Clinically significant new illness in the 1 month before screening
3. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol
4. History of any of the following cardiovascular conditions:

   * Myocardial infarction (diagnosed by cardiac enzyme[s] and/or diagnostic ECG), CVA, TIA or RIND within 6 months of screening
   * Cardiac arrhythmia requiring initiation of new medical or surgical treatment within 6 months of screening (stable medical therapy for > 6 months, pacemakers and/or defibrillators implanted > 6 months prior to screening are acceptable)
   * Unstable angina
5. Surgically implanted portacaval shunts are excluded with the following exception: transjugular intrahepatic portosystemic shunts (TIPS) will be allowed if placed no less than 3 months prior to dosing
6. Malignancy within 2 years of the screening visit (except basal cell or squamous cell carcinoma with clean surgical margins)
7. Initiation of a new prescription medication within 1 month prior to screening.
8. Recent history (within 3 months prior to the screening visit) of alcohol or drug/solvent abuse or a positive screen for drugs of abuse at screening.
9. Use of SSRI's, SNRI's, and other medications must meet the required washout periods.
10. Participated in any clinical study with an investigational drug, biologic, or device within 1 month prior to dosing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the pharmacokinetic properties of lorcaserin in subjects with mild or moderate hepatic impairment compared to subjects with normal hepatic function.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of lorcaserin

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States

REFERENCES:
- [Derived] Christopher RJ, Morgan ME, Tang Y, Anderson C, Sanchez M, Shanahan W. Pharmacokinetics and Tolerability of Lorcaserin in Special Populations: Elderly Patients and Patients with Renal or Hepatic Impairment. Clin Ther. 2017 Apr;39(4):837-848.e7. doi: 10.1016/j.clinthera.2017.03.004. Epub 2017 Mar 30. PMID 28365033